CLINICAL TRIAL: NCT01897168
Title: Bone Mineral Content in Healthy Children
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 135180
Record Dates: First submitted 2013-03-27; First posted 2013-07-11 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine may be collected from study participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No grouping
  Interventions: Device: No intervention

INTERVENTIONS:
Device: No intervention

SUMMARY:
The primary purpose of this study is to determine the effects of early diet on bone health.

ELIGIBILITY:
Inclusion Criteria:

* Current or past participation in the Beginnings study (IRB#07180)
* Age 5-7 years

Exclusion Criteria:

* Growth or bone disorders
* Non-removal metal on participant
* Any other conditions that may affect the outcome of interest as determined by the PI.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Bone health assessed by pQCT and DXA | 5-7 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ran Chen, Ph.D., Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States